CLINICAL TRIAL: NCT00496405
Title: The Role of Unilateral Intravitreal Bevacizumab (Avastin), for the Treatment of Bilateral Diabetic Macular Edema: a Pilot Study.
Brief Title: Unilateral Bevacizumab for Bilateral Diabetic Macular Edema
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APEC
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Macular Edema; Diabetic Retinopathy
Keywords: Vascular endothelial growth factor.; Retinal Thickness; Diabetic Macular Edema; Optical Coherent Tomography
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bevacizumab

SUMMARY:
The endothelial growth factor (VEGF), has been implied in the genesis of diverse Neovascular disease. In the industrialized and developing countries, the main cause of blindness is the diabetic retinopathy. Bevacizumab (Avastin, genentech, Inc., San Francisco, California, the USA) is a drug.In the last years its use "off-label", in ophthalmology field, has become popular. This is due to its proven safeness and effectiveness for the treatment of diverse ocular diseases. A lot has been speculated about the systemic absorption of Bevacizumab. It is for that reason that the objective of this study is the systematic and random revision of the fellows eyes, of the patients programmed for the intravitreal administration of Bevacizumab, with bilateral macular edema. In such a way that the therapeutic value in the fellow eye of bevacizumab can be determined

DETAILED DESCRIPTION:
Introduction:

The endothelial growth factor (VEGF), was identified for the first time in the liquid of ascitis in Guinean pigs (6,7). It is a dimeric glycoprotein, naturally expressed in epithelial and tumor cells (1). It's over expression during retinal hypoxia (9), has been implied in the genesis of diverse Neovascular diseases (2,4,8,9,19). The activation of the VEGF pathway promotes endothelial cells growth, increases the growth, migration and survival of the existing vasculature and produces the differentiation and migration of the endothelial mother cells from the bone marrow towards the general circulation (4). It is also a vasculature permeability factor, because it favors the formation of vascular fenestrations, which produces the exit of liquid and protein deposit in the tissue interstice, favoring the formation of macular edema and neovascularisation (3,8-10).

Its activity is mediated by two tyrosine related receptors of high affinity: the VEGFR 1 (FLT-1) and VEGFR 2 (FLT-2) (1,9). The FLT-1 promotes the cellular proliferation whereas the FLT-2 the migration and the interaction between cells and extracellular matrix(4,5,10)

In the industrialized and developing countries, the main cause of blindness is the diabetic retinopathy (9). Followed close in the United States and Europe by Age related Macular Degeneration (10). The most frequent cause of loss of vision in diabetic retinopathy is macular edema (7). Its incidence is between 13.9 to 25.4% (15). It is characterized by the accumulation of intraretinal liquid at level of the outer plexiform and internal nuclear layers, with the subsequent thickening of the macula (13,15). The diabetic macular Edema is associated to high levels of VEGF in the vitreous (7,8,9). At the moment, the gold standard in the treatment of the proliferative retinopathy is the laser photocoagulation(9). The photocoagulation of the macular area for the treatment of diffuse or focal edema, produces a 50% decrease risk of severe visual loss. Nevertheless the long-term prognosis continues being poor (15).

The Optical Coherent Tomography (OCT) is a relative new, noninvasive technique (12,14), based in low frequency interferometry phenomenon. It is able to provide cross-sectional retinal images (11,12,15,17). It has a resolution of 10-15mm. thanks to that, it is also able to quantitatively measure macular thickness (10,12,14,15,17). The measurements obtained with this system are highly reproducible and they correlated with patient visual acuity (7,11,14,16,17,19). It is very useful when evaluating the vitreous-retinal interface and retinal adherences(11). In the macular edema OCT displays low reflectivity images with increase of retinal thickness(11,13). The classification of macular edema by OCT images, proposed by Dr. Otani (16) and modified by Kang (15) consists of 4 types: Type 1, thickening of the fovea with homogenous optical reflectivity in the entire retina. Type 2, thickening of the retina with noticeable diminution of the optical reflectivity in the external layers of the retina. Type 3, thickening of the fovea with accumulation of subfoveal liquid and a defined border of detached retina. Type 3A without foveal traction, 3B with foveal traction (15).

Bevacizumab (Avastin, genentech , Inc., San Francisco, California, the USA) is a drug, approved by the FDA for the treatment of the metastatic colorectal cancer(2). It consists of a humanized monoclonal antibody that binds all active forms of VEGF (3,18,19), blocking the activity of its two receptors (4). In the last years its use "off-label", in ophthalmology field, has become popular. This is due to its proven safeness and effectiveness for the treatment of diverse ocular diseases (2-4,7,20). Within the ophthalmic pathologies that have been treated successfully with the Intravitreal administration of Bevacizumab, we can mention different Neovascular pathologies (diabetic Retinopathy (9,18), age related macular degeneration(2,4,18)) and pathologies that alter the vascular permeability (macular edema (4,7), Central and branch retinal vein occlusion (3,8,20), central serous choroidopathy). In all of them , treatment responses is characterized by an improvement of the visual acuity, decrease of macular thickness and improvement of the angiographic patterns (8,10). The potential complications of the use of Bevacizumab are the severe thromboembolic event, arterial hypertension (18), epistaxis, proteinuria,hemoptysis, alteration in wound healing and gastrointestinal bleed (4,10).

Exposition of the Problem:

A lot has been speculated about the systemic absorption of Bevacizumab. In a study at the Bascom Palmer Eye Institute, doctors Rosenfeld, Puliafito et al demonstrated the effectiveness of the systemic application of Bevacizumab for the treatment of the age related macular degeneration applying dose of 5mg/Kg. thus Demonstrating, the passage of the molecule from the systemic circulation to specific tissue in both eyes(10). Recently, doctor Bakri and her team at Mayo Clinic in Rochester, Minnesota, establish that a small portion of intravitreal bevacizumab is able to pass to the systemic circulation (1.6% of the injected dose) obtaining detectable concentrations in the vitreous of the fellow eye (11.17ng/ml) at week number 4 after the treatment (21). In the same way, we have cases in our hospital, reported like anecdotal cases, of Bevacizumab application in one eye and improvement of the base pathology in the fellow eye.

It is for that reason that the objective of this study is the systematic and random revision of the fellows eyes, of the patients programmed for the intravitreal administration of Bevacizumab, with bilateral macular edema. In such a way that the therapeutic value of the small concentrations reached in the vitreous of the fellow eye of bevacizumab can be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patient greater of 30 years old, with bilateral diffuse diabetic macular edema, with any degree of diabetic retinopathy that has been programmed for Bevacizumab intravitreal administration in one of both eyes.
* Bilateral macular Thickening, measured by OCT of 225mm or bigger.
* Pupil dilatation greater than 5mm.
* Patient with no previous treatment for diabetic macular edema.

Exclusion Criteria:

* Focal diabetic macular edema or macular edema of different etiology, besides diabetes. (uveitis, pseudophakic patients, vitreous-retinal traction, CRVO, BRVO, CSC).
* Macular edema 3B patter, measured by OCT, according to the macular edema classification.
* Medical history of severe thromboembolic events, uncontrolled arterial hypertension, transitory ischemic attacks, cardiac stroke, acute cerebral vascular event.
* Pregnant women or breast feeding women
* Know allergy to Bevacizumab

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-04; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Retinal thickness | Interventional

SECONDARY OUTCOMES:
Best corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Raul Velez-Montoya, MD, Principal Investigator — Asociación para Evitar la Ceguera en Mexico
Locations (1):
- Asociación para Evitar la Ceguera en Mexico, Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Velez-Montoya R, Fromow-Guerra J, Burgos O, Landers MB 3rd, Morales-Caton V, Quiroz-Mercado H. The effect of unilateral intravitreal bevacizumab (avastin), in the treatment of diffuse bilateral diabetic macular edema: a pilot study. Retina. 2009 Jan;29(1):20-6. doi: 10.1097/IAE.0b013e318186c64e. PMID 18784623